CLINICAL TRIAL: NCT01960387
Title: A Phase II Study of Clofarabine and Cytarabine for Patients With Newly Diagnosed Acute Myeloid Leukemia Who Have Persistent Disease After Treatment With an Anthracycline and Cytarabine
Brief Title: Phase II Clofarabine and Cytarabine for Newly Diagnosed Acute Myeloid Leukemia
Acronym: UPCI 13-066
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: lack of accrual
Sponsor: University of Pittsburgh (Other)
Responsible Party: Principal Investigator, Michael Boyiadzis, Principal Investigator, University of Pittsburgh
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UPCI 13-066
Record Dates: First submitted 2013-10-07; First posted 2013-10-10 (Estimated); Results first posted 2016-08-02 (Estimated); Last update posted 2016-08-02 (Estimated); Status verified 2016-06

CONDITIONS: Acute Myeloid Leukemia
Keywords: AML; clofarabine; cytarabine; persistent AML; induction therapy
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Clofarabine; Antimetabolites; Purine Nucleosides; Cytarabine; pyrimidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Clofarabine and Cytarabine (Experimental): Clofarabine will be administered as a 1-hour (range: 1 hour minimum to 2 hours maximum) intravenous infusion at a dose of 40mg/m2 daily on days 1 through 5. Cytarabine at a dose of 1g/m2 daily will then be given as a 2-hour intravenous infusion, starting 3 hours after the completion of clofarabine administration on days 1 through 5.
  Interventions: Drug: Clofarabine; Drug: Cytarabine

INTERVENTIONS:
Drug: Clofarabine — Clofarabine will be administered as a 1-hour (range: 1 hour minimum to 2 hours maximum) intravenous infusion at a dose of 40mg/m2 daily on days 1 through 5.
  Other Names: Clolar; antimetabolite; Purine nucleoside analog
Drug: Cytarabine — Cytarabine at a dose of 1g/m2 daily will be given as a 2-hour intravenous infusion, starting 3 hours after the completion of clofarabine administration on days 1 through 5.
  Other Names: Cytosine arabinoside; antimetabolite; Pyrimidine analog

SUMMARY:
The combination of clofarabine and cytarabine is an effective and reasonably well-tolerated treatment regimen in patients with either relapsed/refractory or newly diagnosed AML. For this prospective study, we propose the use of clofarabine and cytarabine for second course induction therapy for patients with persistent AML after treatment with an anthracycline and cytarabine.

DETAILED DESCRIPTION:
The primary objective of this prospective study is to evaluate the efficacy (i.e., complete response rate) of clofarabine and cytarabine as second course therapy for the treatment of AML. The secondary objectives are to assess the treatment-related toxicities, to determine the overall and relapse-free survival for patients with AML who are treated with this regimen, and to evaluate potential factors that are predictive of response.

The investigational nature and objective of this study, the procedures involved and their associated risks, potential benefits, and potential alternative therapies will be explained to the patient, and a signed informed consent document will be obtained. Once consented, eligible patients will be treated by the acute leukemia service on the University of Pittsburgh Cancer Institute inpatient unit.

Prior to the start of chemotherapy, patients will receive dexamethasone and ondansetron as pre-medication. Clofarabine will then be administered as intravenous infusion on days 1 through 5. Patients will be monitored closely with vital signs. Cytarabine will then be given as intravenous infusion, starting 3 (maximum of 4) hours after the completion of clofarabine administration on days 1 through 5.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with newly diagnosed AML based on the World Health Organization classification who have persistent disease after their first course treatment with an anthracycline and cytarabine
2. Able to understand and have the ability to provide written informed consent
3. Patients over 18 years of age
4. Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1, or 2
5. Left ventricular ejection fraction (LVEF) ≥ 50%
6. Negative urine pregnancy test for all females
7. All subjects must agree to use an effective method of contraception while receiving the study drugs

Exclusion Criteria:

1. Diagnosis of acute promyelocytic leukemia
2. Relapsed AML
3. Prior use of clofarabine
4. Previous allogeneic or autologous hematopoietic cell transplantation
5. Impaired liver function (serum total bilirubin > 2.0 mg/dL, alanine aminotransferase and aspartate aminotransferase ≥ 4 x the upper limit of normal)
6. Impaired renal function (serum creatinine ≥ 2.0 mg/dL)
7. Uncontrolled or life-threatening infection that is not responding to antimicrobial therapy
8. History of a psychiatric disorder which may compromise compliance with the protocol or which does not allow for appropriate informed consent
9. Concurrent active malignancy; exceptions include patients who have been disease free for 5 years, patients with a history of completely resected non-melanoma skin cancer or successfully treated in situ carcinoma, or patients with another malignancy that is indolent or definitively treated
10. Evidence of severe or uncontrolled systemic diseases (e.g., unstable or uncompensated respiratory or cardiac disease)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2013-10; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Boyiadzis, M.D., M.H.Sc, Principal Investigator — University of Pittsburgh
Locations (1):
- UPMC Hillman Cancer Center, Pittsburgh, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Clofarabine (40mg/m^2/Day) + Cytarabine (1g/m^2/Day): Patients with newly diagnosed Acute Myeloid Leukemia who received clofarabine administered as a 1-2 hour intravenous infusion at a dose of 40mg/m^2 daily plus cytarabine at a dose of 1g/m^2 daily, 2-4 hours maximum intravenous infusion starting 3-4 hours post completion of clofarabine administration on days 1 through 5.
Period: Overall Study
Arm/Group | Clofarabine (40mg/m^2/Day) + Cytarabine (1g/m^2/Day)
Started | 2
Completed | 2
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Patients with newly diagnosed AML based on the WHO classification, who have persistent disease after their first course treatment with an anthracycline and cytarabine.
Arm/Group | Clofarabine (40mg/m^2/Day) + Cytarabine (1g/m^2/Day)
Number analyzed (Participants) | 2
Age, Continuous [Mean (Full Range); unit: years] | 55 [50 to 60]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 2

OUTCOME MEASURES:

1. Primary Outcome: Complete Clinical Response
Description: Number of patients with newly diagnosed Acute Myeloid Leukemia who achieved Complete Response to therapy as determined by bone marrow biopsy evaluation. A CR designation required that the patient achieved a morphologic leukemia-free state and an absolute neutrophil count greater than or equal to 1.0 x 10^9/l, a platelet count greater than or equal to 100 x 10^9/l, and no evidence of extramedullary disease.
Time Frame: Between 14 and 28 days from start of study treatment
Population: Newly diagnosed Acute Myeloid Leukemia patients who received clofarabine (1-2 hour intravenous infusion of 40mg/m2 daily dose) plus cytarabine (2-4 hours maximum intravenous infusion of 1g/m2 daily dose) starting 3-4 hours post completion of clofarabine administration on days 1 through 5, who were evaluable for response by bone marrow biopsy.
Measure: Number; unit: participants
Groups:
- Clofarabine (40mg/m^2/Day) + Cytarabine (1g/m^2/Day): Clofarabine administered as a 1-2 hour intravenous infusion at a dose of 40mg/m^2 daily plus Cytarabine at a dose of 1g/m^2 daily, 2-4 hours maximum intravenous infusion starting 3-4 hours post completion of clofarabine administration on days 1 through 5.
Arm/Group | Clofarabine (40mg/m^2/Day) + Cytarabine (1g/m^2/Day)
Number analyzed (Participants) | 2
participants | 2

2. Secondary Outcome: Overall Survival
Description: Number of months of survival for newly diagnosed Acute Myeloid Leukemia patients treated with Clofarabine (40mg/m^2/Day) + Cytarabine (1g/m^2/Day).
Time Frame: Up to 24 months
Population: Results data are not available due to low/insufficient subject accrual from early [trial] termination.
Arm/Group | Clofarabine (40mg/m^2/Day) + Cytarabine (1g/m^2/Day)
Number analyzed (Participants) | 0

3. Secondary Outcome: Relapse Free Survival
Description: Number of months of relapse free survival for newly diagnosed Acute Myeloid Leukemia patients treated with Clofarabine (40mg/m^2/Day) + Cytarabine (1g/m^2/Day).
Time Frame: Up to 24 months
Population: Results data are not available due to low/insufficient subject accrual from early [trial] termination.
Arm/Group | Clofarabine (40mg/m^2/Day) + Cytarabine (1g/m^2/Day)
Number analyzed (Participants) | 0

4. Secondary Outcome: Predictive Factors for Response to Treatment.
Description: Evaluation of potential factors that are predictive of clinical response in newly diagnosed Acute Myeloid Leukemia patients treated with Clofarabine (40mg/m^2/Day) + Cytarabine (1g/m^2/Day).
Time Frame: Up to 1 year
Population: Results data are not available due to low/insufficient subject accrual from early [trial] termination.
Arm/Group | Clofarabine (40mg/m^2/Day) + Cytarabine (1g/m^2/Day)
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Groups:
- Clofarabine (40mg/m2/Day) + Cytarabine (1g/m2/Day): Patients with Newly Diagnosed Acute Myeloid Leukemia who received clofarabine administered as a 1-2 hour intravenous infusion at a dose of 40mg/m2 daily plus cytarabine at a dose of 1g/m2 daily, 2-4 hours maximum intravenous infusion starting 3-4 hours post completion of clofarabine administration, on days 1 through 5.
Arm/Group | Clofarabine (40mg/m2/Day) + Cytarabine (1g/m2/Day)
Serious Adverse Events (participants affected / at risk) | 1/2
Other Adverse Events (participants affected / at risk) | 0/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Clofarabine (40mg/m2/Day) + Cytarabine (1g/m2/Day) (N=2)
Febrile neutropenia (Blood and lymphatic system disorders) | 1
Lung infection (Infections and infestations) | 1

LIMITATIONS AND CAVEATS:
Results data is not available for Overall Survival, Relapse-free Survival, or assessment of potential predictive factors for response to treatment, due to early termination leading to small numbers of subjects analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes